CLINICAL TRIAL: NCT01713764
Title: A Pilot Study of the Effects of Diet and Behavioral Interventions on Health in Diabetics
Acronym: SUCCEED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-09549
Record Dates: First submitted 2012-08-24; First posted 2012-10-25 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Type II
Keywords: diabetes; obesity; mindful eating; positive affect; low carbohydrate; diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity | interventions — Diet, Carbohydrate-Restricted; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Carbohydrate Diet (Experimental): Participants will be instructed to follow a low carbohydrate diet: carbohydrate intake 10-50 grams a day not including fiber. Foods permitted include: meats, poultry, fish, eggs, cheese, cream, some nuts and seeds, green leafy vegetables, and most other non-starchy vegetables. Because most individuals self-limit caloric intake, no calorie restriction will be recommended.
  Participants will also be taught information about mindfulness and positive affect practices. The mindfulness-based curriculum will focus on the following elements: training on topics such as mindful meditation, mindful eating, awareness of fullness and hunger signals, and taste satiety. The positive emotion curriculum will include: training on topics such as noticing and savoring positive events, gratitude, positive reappraisal, personal strengths, attainable goals, and acts of kindness.
  Interventions: Behavioral: Low Carbohydrate Diet; Behavioral: Mindfulness and Positive Affect Skills
- American Diabetes Association Diet (Active Comparator): Participants in the American Diabetes Association (ADA) diet group will receive standard ADA advice. The diet includes high-fiber foods (such as vegetables, fruits, whole grains, and legumes), low-fat dairy products, fresh fish, and foods low in saturated fat.
  Participants will also be taught information about mindfulness and positive affect practices. The mindfulness-based curriculum will focus on the following elements: training on topics such as mindful meditation, mindful eating, awareness of fullness and hunger signals, and taste satiety. The positive emotion curriculum will include: training on topics such as noticing and savoring positive events, gratitude, positive reappraisal, personal strengths, attainable goals, and acts of kindness.
  Interventions: Behavioral: American Diabetes Association Diet; Behavioral: Mindfulness and Positive Affect Skills

INTERVENTIONS:
Behavioral: Low Carbohydrate Diet
  Arms: Low Carbohydrate Diet
Behavioral: American Diabetes Association Diet
  Arms: American Diabetes Association Diet
Behavioral: Mindfulness and Positive Affect Skills

SUMMARY:
The study is a small pilot, designed to provide data regarding the feasibility and acceptability of conducting such a study on a larger scale. The present study is a randomized controlled clinical trial comparing two mindfulness-based lifestyle modification programs to help people manage diabetes and lose weight, one using on a low-carbohydrate diet (LC) and the other using a moderate-carbohydrate diet promoted by the American Diabetes Association (ADA). Intervention content will include information about nutrition (carbohydrate restriction or American Diabetes Association recommended diet) and emotion regulation and mindful eating strategies.

DETAILED DESCRIPTION:
Approximately 40 individuals with Type II diabetes or prediabetes will be randomized in a 1:1 ratio to treatment groups. Groups will meet for 12 weekly sessions, then approximately biweekly for 3 sessions, for a total of 15 1.5-2 hour sessions over 4.5 months. Participants will be evaluated at 0, 1 month, 3 months, and 6 months. Our outcome of interest is HbA1c (glycated hemoglobin, a measure indicative of blood glucose levels and tied to diabetes severity).

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, Type 2.
* HgbA1c > 6.0% at screening. This is to confirm the diabetes diagnosis.
* Aged 18 years old and older
* BMI 25 and above.

Exclusion Criteria:

* Condition that will make it difficult for participation. Such as:

  * cancer
  * liver failure
  * unstable coronary artery disease
  * severe emphysema
  * bulimia or strong history of bulimia
  * vegan
* Laboratory evidence of organ dysfunction

  * Abnormal kidney function (serum creatinine)
  * thyroid stimulating hormone out of normal range
* Previous use or new changes in medications that can interfere with the measures used in the study:

  * current use of insulin and no immediate plans to start or increase diabetic mediations.
  * more than 3 oral hypoglycemic medications.
  * use of systemic (oral or IV) corticosteroids in the 6 months prior
  * severe autoimmune disorders
  * initiation of psychiatric medications in past 2 months.
* Weight loss confounds

  * Current use of weight loss medications or supplements.
  * History of or planned weight loss surgery.
* Other

  * Pregnant or planning to get pregnant in the next year, breastfeeding, less than 6 months post-partum.
  * Unable or unwilling to do home glucose monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Change from baseline to 3 months
  We test whether Hemoglobin A1c changes from pre-intervention to 3 months. The key outcome measure will compare the two diet groups, but we will also assess whether statistically significant changes occur within groups from pre-intervention to 3 months.

SECONDARY OUTCOMES:
Hemoglobin A1c | Change from baseline to 6 months
  We test whether Hemoglobin A1c changes from pre-intervention to 6 months. The key outcome measure will compare the two diet groups, but we will also assess whether statistically significant changes occur within groups from pre-intervention to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M Hecht, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

REFERENCES:
- [Derived] Saslow LR, Kim S, Daubenmier JJ, Moskowitz JT, Phinney SD, Goldman V, Murphy EJ, Cox RM, Moran P, Hecht FM. A randomized pilot trial of a moderate carbohydrate diet compared to a very low carbohydrate diet in overweight or obese individuals with type 2 diabetes mellitus or prediabetes. PLoS One. 2014 Apr 9;9(4):e91027. doi: 10.1371/journal.pone.0091027. eCollection 2014. PMID 24717684